CLINICAL TRIAL: NCT03685500
Title: Phase IV, Open Label, Randomized, Clinical Trial to Evaluate the Reversibility of Abacavir/Lamivudine/Dolutegravir CNS-Related Neurotoxicity After Switching to Tenofovir Alafenamide/Emtricitabine/Darunavir/Cobicistat
Brief Title: A Clinical Trial to Evaluate the Reversibility of Abacavir/Lamivudine/Dolutegravir CNS-Related Neurotoxicity After Switching to Tenofovir/Alafenamide/Emtricitabine/Darunavir/Cobicistat (TAF/FTC/DRV/c)
Acronym: DETOX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Collaborators: Janssen-Cilag, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GESIDA 10418
Record Dates: First submitted 2018-09-08; First posted 2018-09-26 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — symtuza

STUDY DESIGN:
Intervention Model Description: A phase IV, multicentre, randomised, open-label, pilot clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Patients who postpone switching from ABC/3TC/DTG to Symtuza® (TAF/FTC/DRV/c) four weeks
  Interventions: Drug: ABC/3TC/DTG + Symtuza® (TAF/FTC/DRV/c)
- Arm 2 (Experimental): Patients who switch from ABC/3TC/DTG to Symtuza® (TAF/FTC/DRV/c) during the baseline visit
  Interventions: Drug: Symtuza® (TAF/FTC/DRV/c)

INTERVENTIONS:
Drug: Symtuza® (TAF/FTC/DRV/c) — Treatment with TAF/FTC/DRV/c during 8 weeks since randomized
  Arms: Arm 2
Drug: ABC/3TC/DTG + Symtuza® (TAF/FTC/DRV/c) — Patients continuing on treatment with DTG/3TC/ABC after the randomization for 4 weeks, and then switch to TAF/FTC/DRV/c for 8 weeks
  Arms: Arm 1

SUMMARY:
A phase IV, multicentre, randomised, open-label, pilot clinical trial to evaluate the Reversibility of abacavir/lamivudine/dolutegravir ( ABC/3TC/DTG) CNS-Related Neurotoxicity After Switching to tenofovir alafenamide/emtricitabine/darunavir/cobicistat (TAF/FTC/DRV/c)

DETAILED DESCRIPTION:
The investigators estimate that 55 participants will need to be included per group, 110 patients in total, to demonstrate the benefit of switching ABC/3TC/DTG to TAF/FTC/DRV/c

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age diagnosed with HIV using conventional serology techniques.
* Current antiretroviral therapy with ABC/3TC/DTG for at least 4 weeks.
* HIV viral load < 50 copies/mL for at least 24 weeks prior to signing the consent form (confirmed by two assays at least 12 weeks apart with viremia < 50 copies/mL between both). If the patient has a recent routine blood test available (≤ 4 weeks) that includes determining HIV viral load, these results may be used for the screening visit. If this test is not available, or the test is more than four weeks old, viral load will be determined on the day of screening in order to confirm that the patient meets this criterion.
* A positive screening test for sleep disorders detected using the sleep quality index (Pittsburgh ).

Exclusion Criteria:

* Determination of at least one HIV viral load ≥ 50 copies/mL in the last 12 weeks.
* Allergy, intolerance or existence of resistance mutations to any of the components of TAF/FTC/DRV/c.
* History of active CNS infections.
* Active psychosis, major depression with psychotic symptoms or autolytic ideation.
* Dementia or mental retardation.
* Drug use with a diagnosis of abuse or dependence according to DSM-5 criteria.
* Illnesses that may interfere with the study procedures.
* Inability to complete any of the study procedures.
* Pregnant or nursing women, as well as women of childbearing age who do not agree to use an adequate birth control method.
* Patient with documented intolerance or hypersensitivity to the study medication, or who has a contraindication to use it, according to the technical data sheet

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who self-reported insomnia, between HIV-suppressed patients who continue ABC/3TC/DTG and those who switched to TAF/FTC/DRV/c | week 4
  To compare, between the two arms of the study, changes in the percentage and in the severity of neuropsychiatric symptoms compiled using the Pittsburgh sleep quality index (PSQI). The PSQI contains 19 questions in total. These questions are combined to form seven areas with their corresponding score, each of which shows a range between 0 and 3 points. In all cases, a score of "0" indicates ease, while a score of 3 indicates medium difficulty, within their respective area. The score of the seven areas is finally added for a global score, which ranges from 0 to 21 points. "0" indicates ease of sleep and "21" severe difficulty in all areas

SECONDARY OUTCOMES:
Changes in the severity of neuropsychiatric symptoms, between HIV-suppressed patients who continue ABC/3TC/DTG and those who switched to TAF/FTC/DRV/c | week 4
  To compare, between the two arms of the study, changes in the percentage and in the severity of neuropsychiatric symptoms compiled using the ACTG adverse effects scale. Researchers will specifically ask the patient about eleven adverse effects at each visit. Each adverse effect will be documented and graduated, according to the criteria established in the "AIDS Clinical Trials Group (ACTG) Division of AIDS scale (2014)". Each adverse effect will be assigned a score between 0 and 3 points. The Score will include the individual scores for each of the eleven adverse effects collected, as well as the sum of all the individual scores presented by each patient at each study visit
Changes in the severity of neuropsychiatric symptoms, between HIV-suppressed patients who continue ABC/3TC/DTG and those who switched to TAF/FTC/DRV/c | week 4
  To compare, between the two arms of the study, changes in the percentage and in the severity of neuropsychiatric symptoms compiled using the hospital anxiety and depression scale. The scale includes 14 questions to evaluate the presence of depressive symptoms during the last week. Each question contains four answers with score between 0 and 3 points. To obtain the results of the questionnaire, the researcher must add the score obtained in the 7 questions of anxiety on the one hand and the 7 questions of depression on the other
Changes in the severity of neuropsychiatric symptoms potentially associated with the use of ABC/3TC/DTG after switching to TAF/FTC/DRV/c | Week 4 and 8 after switching to TAF/FTC/DRV/c
  To evaluate the change in the percentage and in the severity of neuropsychiatric symptoms compiled using the ACTG adverse effects scale
Changes in the severity of neuropsychiatric symptoms potentially associated with the use of ABC/3TC/DTG after switching to TAF/FTC/DRV/c | Week 4 and 8 after switching to TAF/FTC/DRV/c
  To evaluate the change in the percentage and in the severity of neuropsychiatric symptoms compiled using the Pittsburg sleep quality index (PSQI)
Proportion and severity of neuropsychiatric symptoms potentially associated with the use of ABC/3TC/DTG after switching to TAF/FTC/DRV/c | Week 4 and 8 after switching to TAF/FTC/DRV/c
  To evaluate the change in the percentage and in the severity of neuropsychiatric symptoms compiled using the hospital anxiety and depression scale.
Percentage of virologic failure after switching antiretroviral therapy from ABC/3TC/DTG to TAF/FTC/DRV/c | Week 8 after switching to TAF/FTC/DRV/c
  Virologic failure is defined as the presence of two consecutive HIV viral loads ≥ 50 copies/mL.

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Univ. 12 de Octubre, Madrid
  - H. Univ. Príncipe de Asturias, Madrid
  - Hospital Fundación Jimenez Diaz, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No